CLINICAL TRIAL: NCT00310765
Title: Pregabalin for the Treatment of Abdominal Pain From Adhesions: Placebo Controlled Trial
Brief Title: Pregabalin for Abdominal Pain From Adhesions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated by the sponsor due to low accrual.
Sponsor: Henry Ford Health System (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ann L. Silverman, DIRECTOR OF GI RESEARCH, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3727
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Pain; Surgical Adhesions
Keywords: abdominal pain; surgical adhesions
MeSH Terms: conditions — Abdominal Pain; Tissue Adhesions | interventions — BID protein, human; Pregabalin

STUDY DESIGN:
Intervention Model Description: Patients were evaluated for the study and were entered into the study if they had documented abdominal adhesions and a daily pain score of 40 mm on a visual assessment scale and 4 on an eleven point Likert scale (0 none and 10 most pain). Patients were randomly assigned to active drug or look alike placebo for 7 weeks followed by an open label phase in which all patients received active drug pregabalin 300 mg daily for 4 weeks measuring pain and sleep scores during each phase of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinding was done to ensure minimum bias. Clinicians were not involved in the randomization process. Patients and clinicians were blinded to the identity of the drug as a look alike placebo was used. The randomization code was was maintained by the research assistant and kept in a locked file cabinet. Separated individuals generated the allocation sequence. The blind was maintained until all the decisions regarding data evaluability were made or in the event of a serious adverse event.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin 150 or 300 mg daily for severe abdominal pain from adhesions (Active Comparator): Patients were randomly assigned to active drug 75-150 mg of pregabalin po BID for 7 weeks followed by a 1 week wash out phase and then were given 150 mg of pregabalin BID for an additional 4 weeks. Daily pain and sleep scores were reported by the patient throughout the study.
  Interventions: Drug: Pregabalin 75 or 150 mg BID for 7 weeks followed by open label pregabalin 150 mg BID for 4 weeks
- Look alike placebo 150 or 300 mg daily for severe abdominal pain from adhesions (Placebo Comparator): Patients were randomly assigned to look alike placebo 75 or 150 mg po BID for 7 weeks followed by a 1 week wash out phase and then were given 150 mg of pregabalin BID for an additional 4 weeks. Daily pain and sleep scores were reported by the patient throughout the study.
  Interventions: Drug: Pregabalin 75 or 150 mg BID for 7 weeks followed by open label pregabalin 150 mg BID for 4 weeks; Drug: Placebo first followed by open label pregabalin

INTERVENTIONS:
Drug: Pregabalin 75 or 150 mg BID for 7 weeks followed by open label pregabalin 150 mg BID for 4 weeks — First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days and treat for 7 weeks. Followed by open label pregabalin for 4 weeks at 150 mg BID
  Other Names: Lyrica
Drug: Placebo first followed by open label pregabalin — Look alike placebo 75 mg po BID and increase to 150 mg BID after 3 days if no improvement for 7 weeks. Open label pregabalin 150 mg BID for last 4 weeks of study.
  Other Names: Look alike placebo followed by open label pregabalin; Lyrica
  Arms: Look alike placebo 150 or 300 mg daily for severe abdominal pain from adhesions

SUMMARY:
The purpose of this study is to evaluate if pregabalin demonstrates significant reduction in abdominal pain from adhesions.

DETAILED DESCRIPTION:
The study will be prospective, double-blinded and randomized. The study will run for 12 weeks. During the first 7 weeks there will be 2 groups in the study with subjects receiving a placebo or the study drug. During the last 4 weeks of the study, all subjects will be offered the study medication, pregabalin. The primary outcome measure will be pain relief documented by a 2-point change on the Likert pain scale with a secondary pain measure of sleep interruption.

ELIGIBILITY:
Inclusion Criteria:

* Must have history of prior surgery and documented adhesions during laparoscopy or open laparotomy within 5 years
* Must have undergone an evaluation to exclude other causes of abdominal pain
* Abdominal pain must be present for greater than three months duration

Exclusion Criteria:

* Patients that are pregnant or breast feeding
* Prior treatment with gabapentin, pregabalin or demonstrated sensitivity to these drugs
* Patients who are immunocompromised
* Patients with significant hepatic or renal insufficiency, or any significant hematologic disorder
* History of illicit alcohol or drug abuse within one year
* Documented serious or unstable medical or psychological condition
* Malignancy within the past 5 years other than in situ squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann L Silverman, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, West Bloomfield, Michigan, United States

REFERENCES:
- [Result] Silverman A, Samuels Q, Gikas H, Nawras A. Pregabalin for the treatment of abdominal adhesion pain: a randomized, double-blind, placebo-controlled trial. Am J Ther. 2012 Nov;19(6):419-28. doi: 10.1097/MJT.0b013e318217a5f5. PMID 22020082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was performed between December 2005 and August 2008. Patients were referred to the gastroenterology clinic if they had documented adhesions in the last 5 years, negative pain evaluation and pain that was thought to be from adhesions.
Pre-assignment Details: After signing consent patients completed a one week baseline pain and sleep evaluation. Patients completed a Short-Form McGill Pain Questionaire during screening and at randomization. Patients had an average daily diary score of at least 4 on the the Likert scale during the baseline week and 5 diary recordings with stable pain medication doses.
Groups:
- Active Drug: 75-150 mg of pregabalin po BID
  Pregabalin : First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg pregabalin and increase to 150 mg po BID if no improvement after 3 days
- Placebo: Placebo 75 or 150 mg po BID
  Pregabalin : 75 mg po BID
  Pregabalin : First 7 weeks 75 or 150 mg of placebo pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days
Period: Placebo Controlled Double Blind
Arm/Group | Active Drug | Placebo
Started | 11 | 7
Completed | 8 | 5
Not Completed | 3 | 2
Period: Open Label
Arm/Group | Active Drug | Placebo
Started | 8 | 5
Completed | 7 | 3
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active Drug: 75-150 mg of pregabalin po BID
  Pregabalin : First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days
- Placebo: Placebo 75 or 150 mg po BID
  Pregabalin : 75 mg po BID
  Pregabalin : First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 16
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.27 (11.73) | 48.85 (16.94) | 46.05 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Absolute Adhesional Abdominal Pain Score Assessed at Baseline Through Week 12 in Patients Treated With Pregabalin 150-300 mg Daily Compared With Patients Given Look Alike Placebo
Description: Patients were randomized to pregabalin or placebo 75 mg twice a day. Patients were allowed to double the dose on day 3 if adequate pain relief was not obtained. Abdominal pain reduction was measured on a Likert scale. A Likert scale assumes the intensity of pain is linear on a continuum from no pain at level 0 to severe pain at level 10. Patients were required to complete a daily dairy recording pain using the Likert 11-point numeric scale. The primary end point was a positive change in the daily pain diary of 2 points from each patient's baseline at weeks 8 after the completion of the blinded study and at week 12 during the open label portion of the study. After 7 weeks all patients are randomized to study drug pregabalin 150 to 300 mg daily for 4 additional weeks after a one week wash out with no medication.
Time Frame: Baseline and week 2 through week 12
Population: The number of patients required per treatment group to achieve greater tha 80% power with alpha=0.05 were based on rates from published articles. The study was terminated early due to low enrollment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients Treated With Placebo: Patients treated with look alike pregabalin placebo 75 or 150 mg BID for seven weeks followed by a week wash out and 150 mg BID of pregabalin
- Patients Treated With Pregabalin: Patients treated with pregabalin 75 or 150 mg po BID
Arm/Group | Patients Treated With Placebo | Patients Treated With Pregabalin
Number analyzed (Participants) | 7 | 11
units on a scale
  baseline pain score | 5.8 (0.96) | 6.15 (0.72)
  week 2 | 5.22 (2.29) | 2.87 (2.28)
  week 3 | 4.64 (1.66) | 1.88 (1.0)
  week 4 | 4.84 (1.28) | 3.31 (2.60)
  week 5 | 4.32 (1.57) | 2.72 (2.05)
  week 6 | 3.88 (1.82) | 2.49 (1.7)
  week 7 | 3.92 (1.76) | 2.53 (2.19)
  week 8 open label with no study medication: number analyzed (Participants) | 3 | 7
  week 8 open label with no study medication | 4.13 (0.51) | 2.46 (2.36)
  week 9 open label: number analyzed (Participants) | 3 | 7
  week 9 open label | 2.21 (0.74) | 2.06 (2.24)
  week 10 open label: number analyzed (Participants) | 3 | 7
  week 10 open label | 2.27 (0.74) | 1.84 (2.13)
  week 11 open label: number analyzed (Participants) | 3 | 7
  week 11 open label | 2.23 (1.55) | 1.46 (2.03)
  week 12 open label: number analyzed (Participants) | 3 | 7
  week 12 open label | 1.13 (1.15) | 1.68 (1.93)
Statistical Analysis 1: Comparison: Patients Treated With Placebo vs Patients Treated With Pregabalin; The number of patients required per treatment group to achieve a >80% power with an alpha=0.05 were based on exact rates from reference articles cited in the paper. Patients were randomly assigned to active drug (pregabalin) or look alike placebo; Test type: Superiority or Other — The group-by-time interaction result from repeated-measure analysis of variance modeling was used to evaluate whether the two study groups differed regarding the pain score change that occurred across each of the two study phases (weeks 0-7 and weeks 7-10). To conform to the analysis of variance assumption of distributional normality, the pain scores were square root transformed before the analysis; p < 0.05, ANOVA; Mean Difference (Net) = 2.0, 95% CI 2-sided [0.0 to 4.0], Standard Deviation 1.5

2. Secondary Outcome: Improved Sleep Scores
Description: Absolute Improvement in Sleep by assessing Mean Daily sleep interference scores as measured weekly starting at baseline and reported weekly through week 12 excluding the first week. This score is an 11 point scale the documents the pain interference in sleep in the preceding 24 hours. 0 is no interference and 10 is pain completely disrupted sleep in the previous 24 hours. During the study patients recorded a daily sleep interference score based on 11 point scale (0-10) with the higher number being the most sleep interference
Time Frame: Baseline and week 2 through week 12
Population: Pregabalin patients received 150mg or 300 mg for seven weeks and placebo patients received a look alike placebo for seven weeks. All patients received open label 300 mg of placebo for 4 weeks after a one week wash out phase at week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Patients received look alike placebo 75 mg or 150 mg BID for 3 days and were able to increase 75 mg placebo to 150 mg placebo BID if no improvement for 7 weeks followed by a 1 week washout period with no study medication. Followed by 4 weeks of active medication 300 mg BID
- Pregabalin: Patients received pregabalin 75 mg BID for 3 days with the ability to increase to 150 mg BID for 7weeks. Then there was a one week period in which no study medication was given followed by 4 weeks in which the participants were given 300 mg of pregabalin BID.
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 7 | 11
units on a scale
  baseline | 4.66 (2.79) | 3.94 (2.22)
  week 2 | 3.4 (3.41) | 2.20 (2.36)
  week 3 | 3.26 (3.11) | 1.60 (1.72)
  week 4 | 3.54 (2.81) | 1.68 (1.78)
  week 5 | 3.06 (2.90) | 1.68 (1.75)
  week 6 | 2.74 (2.60) | 1.55 (1.77)
  week 7 | 3.18 (2.27) | 1.6 (2.09)
  week 8 open label no study medication: number analyzed (Participants) | 3 | 7
  week 8 open label no study medication | 3.30 (1.13) | 1.82 (2.15)
  week 9 open label: number analyzed (Participants) | 3 | 7
  week 9 open label | 1.70 (0.88) | 1.31 (1.84)
  week 10 open label: number analyzed (Participants) | 3 | 7
  week 10 open label | 1.25 (0.98) | 1.37 (1.83)
  week 11 open label: number analyzed (Participants) | 3 | 7
  week 11 open label | 1.18 (0.95) | 1.39 (2.04)
  week 12 open label: number analyzed (Participants) | 3 | 7
  week 12 open label | 0.56 (0.55) | 1.01 (1.43)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; The number of patients required per treatment group to achieve a >80% power with an alpha=0.05 were based on the exact rates from the reference articles cited in the paper; Test type: Superiority or Other — The group-by-time interaction result from repeated-measures analysis of variance modeling was used to evaluate whether the two study groups differed regarding the sleep score change that occurred during the two study phases (weeks 0-7 and weeks 7-11. to conform to the analysis of variance assumption of distributional normality the sleep scores were square root transformed before the analysis; p < 0.05, ANOVA; Mean Difference (Net) = 2.0, 95% CI 2-sided [0.0 to 4.0], Standard Deviation 1.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 5 months. Enrolled patients were scheduled for a minimum of three visits after the first week of treatment at weeks 4,8 and 12 for physical examination, symptom assessment and laboratory studies. Patients were contacted by phone 2 months after completing the study to review general health and adverse events. Deaths and/or adverse events were not monitored/assessed separately between the double-blind and open-label phases in the Active Drug arms.
Groups:
- Active Drug 150 mg Double-blind and 300 mg Open-label: Double-Blind: 75 mg of pregabalin po BID (Weeks1-7) Open-label:150 mg of pregabalin BID (Weeks 8-11)
  Pregabalin : First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days
- Active Drug 300mg Double-blind and 300mg Open-label: Double blink:150 mg of pregabalin BID (Weeks 1-7) Open-label: 150 mg of pregabalin BID (Weeks 8-11)
  Pregabalin : First 7 weeks 75 or 150 mg of pregabalin po BID. Start at 75 mg and increase to 150 mg po BID if no improvement after 3 days
- Placebo (150 mg or 300mg): Double-Blind: Double-blind: Placebo (150 or 300 mg) for weeks 1-7 only.
- Placebo (300 mg Active Drug): Open-label Only: Participants who received placebo during the Double-blind phase had the option to receive pregabalin 150 mg BID during the open-label phase for 4 weeks (Weeks 8-11 only).
Arm/Group | Active Drug 150 mg Double-blind and 300 mg Open-label | Active Drug 300mg Double-blind and 300mg Open-label | Placebo (150 mg or 300mg): Double-Blind | Placebo (300 mg Active Drug): Open-label Only
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 3/6 | 2/7 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug 150 mg Double-blind and 300 mg Open-label (N=5) | Active Drug 300mg Double-blind and 300mg Open-label (N=6) | Placebo (150 mg or 300mg): Double-Blind (N=7) | Placebo (300 mg Active Drug): Open-label Only (N=5)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — 60 yo woman did not disclose a history of alcohol abuse. She attempted suicide with an overdose of pregabalin. History available from emergency Psychiatrist. Patient was hospitalized and refused further follow up.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug 150 mg Double-blind and 300 mg Open-label (N=5) | Active Drug 300mg Double-blind and 300mg Open-label (N=6) | Placebo (150 mg or 300mg): Double-Blind (N=7) | Placebo (300 mg Active Drug): Open-label Only (N=5)
headache and hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0
night sweats (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
drowsiness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dizziness and blurred vision (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hand numbness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastroenteritis and dizziness (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pedal edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Difficult to find patients that met criteria for study entry. Study terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No